CLINICAL TRIAL: NCT06041997
Title: Smartphone Use Restriction as Treatment of Primary Headache: a Randomized Controlled Clinical Trial
Brief Title: Smartphone Use Restriction as Treatment of Primary Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Principal Investigator, Deepti Vibha, Clinical Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSIR-642
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone restriction (Experimental): Patients with headache with history of high smartphone use will be randomized into restriction and no-restriction arm.
  Restriction method:
  In the 'run-in' period of four weeks, the smartphone usage will be assessed in terms of number of overall use. The patients will then be advised to cut down the usage by one-third in terms of usage hours. The compliance will be checked at the time of outcome assessment.
  Interventions: Behavioral: Smartphone restriction
- Control (No Intervention): Comparison:
  In the 'run-in' period of four weeks, the smartphone usage will be assessed in terms of number of overall use. In the non-intervention group only the smartphone usage data will be collected in the study period. The non-smartphone users will be as another control arm.

INTERVENTIONS:
Behavioral: Smartphone restriction — The patients will then be advised to cut down the usage by one-third in terms of usage hours. The compliance will be checked at the time of outcome assessment.
  Arms: Smartphone restriction

SUMMARY:
The goal of this clinical trial is to study smartphone use restriction as a treatment modality in patients of primary headache. The main question[s] it aims to answer are:

1. In patients with primary headache, does restriction of smartphone use lead to reduced consumption of medications (acute, prophylaxis, either or both)?
2. In patients with primary headache, does restriction of smartphone use lead to better responsiveness to medications (acute, prophylaxis, either or both)?
3. Can reduction of smartphone duration be used as a non-pharmacological treatment of primary headache?
4. In patients with primary headache, is the type of smartphone use (phone calls, internet browsing, watching screen) determinant of the severity of headache?
5. Can we make an addiction score to predict which patient should be advised to limit smartphone use based on the above information?
6. In patients with primary headache, does restriction of smartphone use led to improvement in headache severity (frequency, intensity, duration, one of them or all).

The smartphone users may further be classified into low and high smartphone users depending upon the smartphone addiction questionnaire (SAQ) (appendix 1) usage score. SUs with 0-1 score on the SAQ were further grouped into low SUs, and patients with score ≥1 were grouped into high SUs. To create a homogenous group, only patients with high SU will be randomized to standard treatment (Arm C) and intervention group (Arm D).

Participants will be asked about their smartphone usage, and if found eligible, there will be a run-in period of 4 weeks after which they will be randomized to the intervention (smartphone restriction) or comparison group (no restriction recommended)

DETAILED DESCRIPTION:
Study description:

Patients/participants:

1. Patients ≥18 years of age
2. Diagnosis of primary headache as per the ICHD3Beta classification ("ICHD-3 The International Classification of Headache Disorders 3rd Edition" n.d.)
3. Willing and consenting to participate in the study. Patients will be first asked about their smartphone use.

   * If they do not use smartphone, they will be asked if they use any phone at all for calling, and their call durations will be recorded over the run-in and study period.
   * If they do not use any phone, they will fall in the external control group (Arm A).
   * If the patient uses a feature phone, but not a smartphone, he/she will be in another external control group (Arm B). These patients will not be randomized, but will be maintained on routine follow-up.
   * If they use smartphone their use will be recorded over the study period in terms of:

     o Screen use: Social network/testing/gaming/surfing/reading/music/video
   * The smartphone users may further be classified into low and high smartphone users depending upon the smartphone addiction questionnaire (SAQ): usage score. SUs with 0-1 score on the SAQ were further grouped into low SUs, and patients with score ≥1 were grouped into high SUs. To create a homogenous group, only patients with high SU will be randomized to standard treatment (Arm C) and smartphone restriction group (Arm D).

Patients with headache with history of high smartphone use will be randomized into restriction and no-restriction arm.

Restriction method:

In the 'run-in' period of four weeks, the smartphone usage will be assessed in terms of number of overall use. The patients will then be advised to cut down the usage by one-third in terms of usage hours. The compliance will be checked at the time of outcome assessment.

Comparison:

In the non-intervention group only the smartphone usage data will be collected in the study period. The non-smartphone users will be as another control arm.

Outcome:

Primary:

The number of times the patient is using acute pain medications for headache per month, within three months after initiation of study period.

Secondary:

1. The frequency of headache over a period of one month, three months after the initiation of study period in the intervention versus control group.
2. The number of prophylaxis medications being taken three months after the initiation of study period in the intervention versus control group.

Timeline of measuring outcome:

The follow up will be over a period of 20 weeks after screening eligibility and 16 weeks after randomization. The patient will maintain a headache diary in which he/she will enter the number of times they needed to take rescue medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. Diagnosis of primary headache as per the ICHD3Beta classification ("ICHD-3 The International Classification of Headache Disorders 3rd Edition" n.d.)
3. Willing and consenting to participate in the study.

Exclusion Criteria:

* 1. Secondary headaches 2. Not consenting for participation or follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The pill burden for abortive treatment | three months after initiation of study period
  The number of times the patient is using acute pain medications for headache in one month

SECONDARY OUTCOMES:
Headache frequency | One and three months
  The frequency of headache over a period of one month, three months after the initiation of study period in the intervention versus control group.
Number of prophylactic medication | Three months
  The number of prophylaxis medications being taken three months after the initiation of study period in the intervention versus control group.

CONTACTS AND LOCATIONS:
Overall Officials: Deepti Vibha, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Deepti Vibha, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the completion of the publication for six months
Access Criteria: Shared on individual request